CLINICAL TRIAL: NCT01976559
Title: Comparison of Continuous Noninvasive and Invasive Intracranial Pressure Measurement--Celda Infusion Subprotocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeBridge Health (Other)
Collaborators: University Hospital, Umeå (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB 1964; SMST02802 (Other Grant/Funding Number: National Space Biomedical Research Institute SMST02802)
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Hydrocephalus; Shunt Malfunction
Keywords: ICP; Intracranial pressure; Hydrocephalus; Idiopathic normal pressure hydrocephalus; CSF; Cerebrospinal fluid; Noninvasive ICP
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydrocephalus / Shunt Malfunction (Experimental): Patients between the ages of 18-80 years with suspected hydrocephalus, shunt malfunction, or disorders of CSF circulation who are recommended by their doctor based on standard clinical criteria to undergo CSF infusion testing. The interventions include tympanic membrane displacement (TMD) and DPOAE.
  Interventions: Device: Tympanic Membrane Displacement (TMD); Device: DPOAE

INTERVENTIONS:
Device: Tympanic Membrane Displacement (TMD) — The CCFP Analyser has a passive mode and an active mode. When used in active mode, the device generates a tone burst that is transmitted to the ear to elicit contraction of the stapedius muscle. The passive mode requires no stimulus or sound burst.
  For each ICP level during the CSF infusion testing, the active mode will be used. Each condition comprises 13 stimuli of 0.3s duration.
  Other Names: Marchbanks MMS-14 TMD Cerebral Cochlear Fluid Pressure (CCFP) Analyzer
Device: DPOAE — DPOAE measurement uses a clinical acoustic probe to record the ear's response to two simultaneous tones. DPOAE measurements will be made for 13 tones. The total measurement time for each condition is 2-4 minutes.
  Other Names: Distortion Product Otoacoustic Emissions

SUMMARY:
This research is being done to determine the accuracy of two noninvasive methods of measuring the pressure of the spinal fluid, also known as intracranial pressure (ICP).

DETAILED DESCRIPTION:
Recently, astronauts in long-duration spaceflight have been found to have a syndrome consisting of swelling of the optic nerve, impaired vision, and elevated cerebrospinal fluid pressure (also known as intracranial pressure [ICP]) via lumbar puncture (LP), which is similar to the syndrome of idiopathic intracranial hypertension (IIH). In astronauts, this syndrome is called Visual Impairment/Intracranial Pressure (VIIP). It is not possible to perform an LP on astronauts in space. Noninvasive methods of estimating ICP exist but have not been tested against continuous ICP methods in a patient cohort that is physiologically similar to that of astronauts.

The primary objective of this study is to determine the validity, reliability, accuracy, and precision of two noninvasive methods of ICP measurement (tympanic membrane displacement (TMD, Marchbanks Measurements Systems, UK) and distortion product otoacoustic emissions (DPOAE) in comparison to a reference standard, invasive ICP measurement, in human subjects undergoing diagnostic cerebrospinal fluid (CSF) infusion testing.

The two noninvasive methods are based on the responses of the inner ear and middle ear to changes in ICP. The first method is TMD, which measures tiny movements of the ear drum, and the second is DPOAE, which is routinely used for newborn hearing screening.

Adults with hydrocephalus, shunt malfunction, or other disorders of CSF circulation who have been recommended on the basis of standard clinical criteria to have CSF infusion testing are eligible.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of suspected hydrocephalus or shunt malfunction
* CSF infusion testing has been recommended on the basis of standard clinical criteria
* Capable of providing valid signed informed consent
* Normal middle-ear function as determined by tympanometry
* DPOAE meet criteria that are required for the research
* Acoustic stapedial reflex meets criteria that are required for the research
* Subject is willing and able to participate in the study

Exclusion Criteria:

* Subject is pregnant
* Subject lacks decision-making capacity
* Subject is unwilling to participate in the study
* Prior middle-ear disease or surgery, with the exception of tympanostomy tubes that have been removed and are healed
* Participating in the study would significantly delay or interfere with the subject's healthcare
* Subject has excess ear wax that cannot be removed safely and could potentially be pushed onto the ear drum by insertion of the ear plugs needed for the testing
* The TMD or DPOAE do not respond to a change in posture from lying flat to standing up, which means that the anatomic connection between the inner ear and the CSF is absent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Noninvasive ICP | Day 1 (Concurrent with CSF infusion testing)
  Bland-Altman analysis: the difference between the noninvasive ICP and the invasive ICP is plotted against the mean of both the noninvasive and invasive ICP at each ICP level

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Williams, MD, Principal Investigator — Sinai Hospital of Baltimore / LifeBridge Health
Locations (1):
- University of Umea Hospital, Umeå, Sweden